CLINICAL TRIAL: NCT03207308
Title: Using Stable Isotope Techniques to Monitor and Assess the Vitamin A Status of Children Susceptible to Infection in Senegal
Brief Title: Vitamin A Total Body Stores of Senegalese Children in Relation to Their Infectious Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheikh Anta Diop University, Senegal (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RAF6047SEN
Record Dates: First submitted 2017-01-24; First posted 2017-07-02 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Infection; Vitamin A Overdose
Keywords: Vitamin A Status; Retinol Isotope dilution; Total body vitamin A stores; Children; Senegal
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin A supplementation (Experimental): 55 children will receive a Mega-dose of preformed Vitamin A as recommended by the Senegalese Ministry of Health
  Interventions: Dietary Supplement: Vitamin A supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin A supplementation — 200,000 IU of preformed vitamin A

SUMMARY:
Despite economic growth in developing countries, Sub-Saharan Africa still faces food insecurity malnutrition and infections. Micronutrient deficiency and infectious diseases still remain a public health problem and have a negative impact on health and the economy. They are both directly and indirectly responsible for children morbidity and mortality. Due to high level of children mortality (139‰) Vitamin A Supplementation (VAS) program was implemented in Senegal since 1999. A national representative study undertook in 2010 to have biological data on vitamin status and infections, showed that 24.4% of children aged 1-5 y were Vitamin A Deficiency (VAD) and 50.2% were infected. To address VAD issue, large scale oil fortification was launched by government and private industries also fortified bouillon cubes. Furthermore, home fortification is being initiated without evaluation of VAD control strategies existing in the country.

In order to assess the impact of national VAD control strategies in Senegalese children, this study was designed to measure in subsample of rural children aged 3-5 y, the current vitamin A total body stores in relation to their infectious status.

DETAILED DESCRIPTION:
Specifics objectives are:

Assess total body vitamin A stores and hepatic reserves before and after vitamin A supplementation in children aged 3-5 y by deuterated-retinol dilution technique Measure plasma retinol, ferritin and zinc concentrations in children Measure plasma C-reactive protein and alpha 1 glycoprotein concentrations and malaria parasitemia Identify health, socioeconomic and food determinants that can influence children micronutrient status

Study design is longitudinal with repeated measures and will be implemented in rural area. Five months after the passage of Vitamin A Supplementation (VAS) campaign, fifty children (n=50) aged 3-5y will be enrolled in the study (randomized sampling) plus 10% for drop out. The protocol will be explained to the mother and written consent will be obtained from her.

Dietary intake information will be collected using 24 hour recall questionnaire, food frequency questionnaire and infections frequency questionnaire will be submitted to the mother at d-7. Anthropometric measurements (weight and height) of children will be recorded also at d-7.

Subjects will receive doses of labeled vitamin A:

6µmol of D4-Vitamin A, and 6 µmol of D8-Vitamin A per children at d0 and d44 respectively. Blood sampling will be done 3 times during the study: at Baseline (d-7) and 2 weeks after each dose of labeled vitamin A (d14 and d58). The blood will be drawn from children and immediately wrapped on aluminum foil and placed in a cooler while in the field. The blood samples will be transported to the lab and treated under dim light (centrifugate and separation in cryogenic vials). C - reactive protein (CRP) and alpha-1 acid glycoprotein (AGP) will be measured by Elisa method. Serum retinol measurement will be done by HPLC after ethanol hexane extraction with 200 µl of serum and vitamin A total body stores by GC-MS.

Others micronutrient determination will be done as Iron (ferritin by Enzyme Linked Fluorescent Assay (ELFA)) and Zn (Atomic Absorption Spectrophotometer by flame).

Anemia will be assessed by measuring hemoglobin (Hb) in whole blood using a HemoCue system (Hb-301) and malaria parasitemia will be measured using Rapid Diagnostic tests (RDT)

Statistical analyses will be carried out with STATA / SE (Special Edition, Stata Corporation, Texas, USA). The results will be expressed as mean ± standard deviation and percentages. The variables with non Gaussian distributions will undergo a logarithmic transformation and will be expressed in geometric mean ± standard deviation.

The analysis of variance (ANOVA) associated with a posteriori test (Bonferroni) will be used for repeated measures and Student's t test will be used for comparison of means. The Chi² test will be used for percentages comparison.

The relationship between quantitative variables will be assessed with the Pearson correlation coefficient. Multiple and logistic regression will be performed to identify the socio-economic, health and dietary determinants of vitamin A status, evaluate their contributions and their influence on the risk of vitamin A deficiency. For all these statistical analysis, a significance level of 0.05 will be applied.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years, not planning to move from the study area for the duration of the study, and do not have severe illness at the time of enrollment.

Exclusion Criteria:

* severe anaemia, severe acute malnutrition, obesity or clinically defined severe illness, such as dehydration, severe diarrhoea or severe respiratory illness.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Vitamin A status 1 | Within the coming 2 years
  Total body pool size vitamin A (mmol)

SECONDARY OUTCOMES:
Acute infection | Within the coming 2 years
  C-reactive protein (CRP) expressed as mg/L
Chronic infection | Within the coming 2 years
  Acide glycoprotein (AGP) expressed as g/L
Iron status | Within the coming 2 years
  Ferritin expressed as µg/L
Stunting | Within the coming 2 years
  Height for Age Z-score
Wasting | Within the coming 2 years
  Weight for Height Z-score and middle upper arm circumference
Underweight | Within the coming 2 years
  Weight for Age Z-score,
Morbidity | Within the coming 2 years
  Medical history of the child enrolled in the study such as diarrhea, fever, malaria, rashes, measles, respiratory infection, vitamin A supplementation, drug for intestinal de-worming, iron supplementation.
Socioeconomic status | Within the coming 2 years
  Quintile of poverty (obtained by aggregation of socioeconomic informations like household (HH) family size, marital status of the head of the HH, source of drinking water, highest level of education the head of HH, etc.)
Dietary intake | Within the coming 2 years
  24h dietary recall and food consumption frequency
Anemia status | Within the coming 2 years
  Hemoglobin expressed as g/L
Malaria parasitemia | Within the coming 2 years
  Presence or absence of plasmodium falciparum antigens

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Loechl, PhD, Study Director — International Atomic Energy Agency
Locations (1):
- Universite Cheikh Anta Diop, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No